CLINICAL TRIAL: NCT06094127
Title: A Post-market Clinical Follow up Study on Cook Medical Zenith® Alpha Thoracic Endovascular Grafts
Brief Title: Zenith Thoracic Alpha (ZTA) Post-Market Data Collection
Status: Recruiting | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 17-13
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Aortic Aneurysm; Penetrating Aortic Ulcer
Keywords: Aneurysm; Thoracic; Descending; Aorta; Stent-graft
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Penetrating Atherosclerotic Ulcer; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Endovascular aortic treatment — Use of ZTA to treat diseases in the descending thoracic aorta, such as thoracic aortic aneurysm and penetrating aortic ulcer.

SUMMARY:
This study aims to gather real-world clinical data demonstrating the continued safety and performance of the a marketed stent graft (Zenith® Alpha Thoracic Endovascular Graft [ZTA]) and collect longer term follow-up to better understand clinical outcomes associated with the expected lifetime of the device.

DETAILED DESCRIPTION:
Per local regulations, this study includes both retrospective and prospective patients. Patients can be included retrospectively if they are treated with the study device from 01 January 2019 until the study site is eligible for prospective enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treated/was intended to be treated with ZTA according to the clinical practice from Jan 2019 until site initiation
* The patient is willing to participate in the study and provide written informed consent for study participation or express non-objection or give written consent per local requirements prior to data collection of any data from medical records.

Exclusion Criteria:

* A patient treated with a custom-made fenestrated and/or branched endovascular graft in conjunction with ZTA either during the same procedure or in a staged procedure.
* A patient whose follow-up data collection is not possible (e.g. due to living abroad).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with a (ZTA) since January 2019through 1 year follow-up from index placement procedure.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2034-12-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from aneurysm-related mortality | 5 years
  Death related to aneurysm

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Tsilimparis, MD, Principal Investigator — Klinikum der Universitat Munchen
Locations (10):
- France (3):
  - CHU Dijon Bourgogne, Dijon
  - Hopital Marie Lannelongue Groupe Hospitalier Pairs St Joseph, Le Plessis-Robinson
  - Centre Hospitalier Regional Universitaire de Lille, Lille
- Germany (3):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum der LMU München, München
  - St. Franzikus Hospital Munster, Münster
- Italy (2):
  - IRCCS-University Hospital Sant'Orsolo Polyclinic, Bologna
  - IRCCS Ospedale San Raffaele, Milan
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Radboud UMC, Nijmegen